CLINICAL TRIAL: NCT06729957
Title: Addressing Barriers to Care for Substance Use Disorder Trial (Center for Dissemination and Implementation At Stanford, Research Component #3)
Brief Title: Addressing Barriers to Care for Substance Use Disorder Trial
Acronym: ABC-SUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Stanford University (Other)
Responsible Party: Principal Investigator, Joseph Glass, Senior Investigator, Chestnut Health Systems
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2068557T; P50DA054072 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Drug Use Disorders; Alcohol-Related Disorders; Substance Use Disorder (SUD)
Keywords: Implementation Science; Care Navigation; Drug Use Disorders; Quality Improvement; Behavioral Health
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders

STUDY DESIGN:
Intervention Model Description: Care coordinators will be randomized to care navigation arm or services as usual arm at study outset and switch to the opposite arm halfway through the study.
Who Masked: Outcomes Assessor
Masking Description: All study outcomes are extracted from electronic health records and healthcare claims data that cannot be manipulated by the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care Navigation (Experimental): Mental health care coordinators are able to offer and refer patients to a care navigator in addition to offering substance use resources and treatment options as usual.
  Interventions: Behavioral: Care Navigation
- Services as Usual (No Intervention): Mental health care coordinators will continue offering substance use resources and treatment options to patients as usual.

INTERVENTIONS:
Behavioral: Care Navigation — Care navigation is an intervention that seeks to help patients engage in substance use treatment by increasing motivation and reducing barriers to accessing treatment. The care navigator helps the patient engage in the treatment plan established by the mental health care coordinator.
  Arms: Care Navigation

SUMMARY:
The Addressing Barriers to Care for Substance Use Disorder Trial (ABC-SUD) is a cluster-randomized crossover trial, with clinicians (care coordinators) as the unit of randomization.

This study will be conducted in a mental health access center within the Washington region of Kaiser Permanente. As part of usual care, patients contact the mental health access center and speak to a care coordinator to obtain an appointment with or contact information for potential venues to obtain treatment for substance use disorder.

The experimental intervention, Care Navigation, will be evaluated for its potential to increase engagement in substance use disorder treatment among patients who contact the mental health access center. Care Navigation will be delivered by study care navigators, who are distinct from the health system's care coordinators.

DETAILED DESCRIPTION:
The ABC-SUD Trial is a cluster-randomized crossover trial evaluating the effectiveness of care navigation in increasing engagement in substance use disorder treatment. Each care coordinator is randomly assigned to a study arm (services as usual or care navigation) at the beginning of the trial (period 1), and halfway through the trial, switches to the other study arm (period 2). The patient population includes individuals who are seeking substance use treatment and are evaluated by enrolled care coordinators.

During periods in which care coordinators are assigned to the intervention arm, care coordinators offer care navigation to patients and utilize an electronic health record referral tool to refer patients to care navigators. This tool is disabled for care coordinators during the period in which they are assigned to the control arm.

This study will employ an encouragement design, where patients who speak with intervention care coordinators are offered care navigation, but patients choose whether to participate in care navigation. Primary analyses will follow an intent-to-treat principle whereby care coordinators and patients will be analyzed according to the intervention arm to which they are assigned regardless of the subsequent sequence of events.

ELIGIBILITY:
Clinician (Care Coordinator) Inclusion Criteria:

* Conducts assessment and treatment planning visits in the mental health access center
* Has been employed for at least 1 month
* Has completed trainings related to their clinical role in the health system
* Scheduled to conduct assessments

Clinician Exclusion Criteria: None

Patient Inclusion Criteria (eligibility for analyses):

* Visits an enrolled care coordinator during the patient eligibility period
* ≥ 18 years of age at the time of the visit
* Has an assessment and treatment planning visit for SUD with an enrolled care coordinator

Patient Exclusion Criteria:

* Patients who have requested through the health system to opt out of research contact or chart review
* Patients who are not enrolled in Kaiser Permanente insurance, or those only enrolled in Medicaid (anticipated incomplete capture of covariate and/or outcome information)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Engagement in treatment for substance use disorder | 48 days
  Completion of ≥ 3 treatment visits for substance use disorder within 48 days of their assessment visit

SECONDARY OUTCOMES:
Initiation of treatment for substance use disorder | 30 days
  Completion of ≥ 1 treatment visit for substance use disorder within 30 days of their assessment visit

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Glass, PhD, MSW, Principal Investigator — Chestnut Health Systems
Locations (1):
- Kaiser Permanente Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
This study protocol is embedded within a Center of Excellence funded by the National Institute on Drug Abuse. In coordination with other center project components, the study protocol will be submitted for publication to either an addiction or implementation science journal. Additional data (analytic code) can be requested from the Principal Investigator. Participant data will be shared with the prime site as allowed. Analysis files will be constructed from the electronic data and aggregated. No names, addresses, telephone numbers, email addresses, medical record numbers, etc. will be retained in the aggregated files.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Anticipated 1/1/2027-12/31/2030
Access Criteria: Plans for data access will be determined in conjunction with the prime site

REFERENCES:
- [Derived] Matson TE, Navarro MA, Idu A, Bobb JF, Patrick BM, Phillips R, Barrett TD, Rossi FS, Krawczyk N, Doud R, Rogers K, Davis CJ, Caldeiro R, Glass JE. Design of a cluster-randomized, hybrid type 1 effectiveness-implementation trial of a care navigation intervention to increase substance use disorder treatment engagement: study protocol. Addict Sci Clin Pract. 2025 Oct 1;20(1):78. doi: 10.1186/s13722-025-00605-7. PMID 41035041